CLINICAL TRIAL: NCT02438267
Title: Preterm Infants and Nephrocalcinosis: Diagnosis and Pathogenesis
Brief Title: Preterm Infants and Nephrocalcinosis
Acronym: NC
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 66906
Record Dates: First submitted 2015-05-01; First posted 2015-05-08 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2016-06

CONDITIONS: Prematurity; Nephrocalcinosis; Hypercalciuria
MeSH Terms: conditions — Premature Birth; Nephrocalcinosis; Hypercalciuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-NC group: Enrolled subjects who did not have evidence of NC on renal ultrasound
- NC group: Enrolled subjects who did have evidence of NC on renal ultrasound

SUMMARY:
Nephrocalcinosis (NC), defined as calcification of renal tissue, has been reported to occur in 7-41% of premature infants. Causes of NC are likely multi-factorial, and infants born prematurely and with very low birth weight (<1500 gm) seem to be at the highest risk of developing NC. Recent changes in recommendations for nutrition for the preterm infant such as higher intakes of protein, calcium, and vitamin D may also play a factor in the pathogenesis of NC.

Currently, diagnosis of NC often occurs incidentally during ultrasound evaluation for other issues. Because there is no acute symptom or pattern of symptoms in the preterm population associated specifically with NC, it is possible that many cases of NC may not be diagnosed. Presently, it is impractical and costly to screen all infants for NC with renal ultrasound, therefore there is no standard of care regarding screening for NC.

NC may have long-term effects. Studies have shown that preterm infants with NC had shorter kidneys and a lower rate of tubule resorption of phosphorus (TRP) than preterm infants without NC.

This study will analyze weekly urinalysis for all enrolled subjects prospectively and then look at the incidence of NC at discharge of the enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

* Infants whose gestation less than or equal to 32 weeks and/or birth weights less than 1800 gm

Exclusion Criteria:

* Infants with congenital abnormalities of the heart, lung, GI, or kidneys that will affect renal function.

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the newborn intensive care unit.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Urinary calcium to creatinine ratio (UCa/Cr) | 3 months
  Beginning within the first two weeks of life, urine calcium to creatinine ratio (UCa/Cr) will be analyzed weekly through discharge and then correlated to renal ultrasound results done prior to discharge.
Urinary crystals | 3 months
  Beginning within the first two weeks of life, urinalysis for evidence of urinary crystallization will be analyzed weekly through discharge and then correlated to renal ultrasound results done prior to discharge.

SECONDARY OUTCOMES:
Serum Vitamin D levels | 3 months
  Serum vitamin D levels will be analyzed and compared in infants with NC against infants without NC (controls).
Vitamin D intake | 3 months
  Daily vitamin D intake will be recorded from participants' medical records and will be analyzed and compared in infants with NC against infants without NC (controls).
Calcium intake | 3 months
  Daily calcium intakes will be recorded from participants' medical records and will be analyzed and compared in infants with NC against infants without NC (controls).
Protein intake | 3 months
  Daily protein intakes will be recorded from participants' medical records and will be analyzed and compared in infants with NC against infants without NC (controls).
Total bone density per DXA | 3 months
  Whole body bone density per dual energy X-ray absorptiometry (DXA) will be done on all enrolled participants at discharge and will be compared between infants with and without NC.
Tibial bone density per tibial ultrasound | 3 months
  Tibial body bone density per ultrasound will be done on all enrolled participants at discharge and will be compared between infants with and without NC.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Malone-Jenkins, MD, Principal Investigator — University of Utah
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States